CLINICAL TRIAL: NCT03319290
Title: Medical Provider Experience Assessment Healthcare Decisions Post-Testing, Risk Reducing, and Preventative Strategies Using BRCA2 and BRCA2 Genetic Testing
Brief Title: Increase Surveillance for Breast and Ovarian Cancers, Also to Determine Targeted Risk-reducing and Preventative Strategies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1460
Record Dates: First submitted 2017-10-17; First posted 2017-10-24 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hereditary Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: BRCA1 and BRCA2 — Genetic breast and ovarian cancer testing

SUMMARY:
Observational study is to increase surveillance for breast and ovarian cancers, also to determine targeted risk-reducing and preventative strategies.

DETAILED DESCRIPTION:
The general design of this study is collecting data and reviewing the Principal Investigators' (P.I.) Standard Operating Procedures (SOP) on BRCA testing and changes made to their specific SOP.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Medical Practitioner

  * Medical Doctor (MD)
  * Doctor of Osteopathic (DO)
  * Physician Assistant (PA)
  * Advanced Practice Registered Nurse (APRN)
  * Nurse Practitioner (NP)
* Must have a current standard operating procedure that includes obtaining/reviewing medical history and family medical history

Exclusion Criteria:

* Government-funded insurance data cannot be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current standard operating procedures for providers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-17 (Estimated)

PRIMARY OUTCOMES:
Provider Structures and Processes | 36 months
  Plan of Care Changes due to BRCA testing. Provider based observational survey system on the health and well-being of patients and populations

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No